CLINICAL TRIAL: NCT02649998
Title: Comparison of Short-term Efficacy of Furosemide, Isosorbide Dinitrate and Their Combination in Patients With Acute Decompensated Heart Failure: A Randomized Controlled Trial
Brief Title: Short-term Efficacy of Furosemide, Isosorbide Dinitrate and Their Combination in ADHF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Colin Graham, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE.2015.592-T
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Heart Decompensation
Keywords: Fursemide; Isosorbide Dinitrate; Heart Decompensation; Clinical Trials, Randomized; Clinical Efficacy
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Isosorbide Dinitrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Each patient will initially receive a 40 mg bolus of IV furosemide (10 mg/mL) and a 2 mL bolus of IV saline placebo, followed by IV saline placebo 6 mL/h
  Interventions: Drug: Furosemide
- Group 2 (Active Comparator): Each patient will initially receive a bolus of IV saline placebo and a 2 mL bolus of IV isosorbide dinitrate (1 mg/mL), followed by IV isosorbide dinitrate 6 mL/h
  Interventions: Drug: Isosorbide Dinitrate
- Group 3 (Active Comparator): Each patient will initially receive a 40 mg bolus of IV furosemide (10 mg/mL) and a 2 mL bolus of IV isosorbide dinitrate (1 mg/mL), followed by IV isosorbide dinitrate 6 mL/h
  Interventions: Drug: Furosemide; Drug: Isosorbide Dinitrate

INTERVENTIONS:
Drug: Furosemide — Furosemide is the most commonly used medication for treatment of heart failure. It causes a direct vasodilator effect shortly after administration, followed by diuresis induction. However, furosemide also activates both the sympathetic and the renin angiotensin systems, causing a rise in peripheral resistance.
  Other Names: Lasix
  Arms: Group 1; Group 3
Drug: Isosorbide Dinitrate — Isosorbide dinitrate is a vasodilator which is also well-known for treating acute decompensated heart failure. It induces acute venodilatation at low dose and arteries dilation when gradually increasing the dose. The effect peaks 5 min after administration.
  Other Names: Isoket
  Arms: Group 2; Group 3

SUMMARY:
Background:

Acute decompensated heart failure (ADHF) is a common and potentially fatal cause of acute respiratory distress that requires immediate treatment in emergency department. The mortality rates are as high as 20% after discharge. Currently, furosemide is the most commonly used medicine in emergency department for ADHF. Although nitrate was proved to generate similar effect when compared to furosemide, less than 30% of patients received nitrates. This practice happens not only in Hong Kong, but also all around the world. Moreover, there is limited evidence to support a difference in ADHF patients receiving intravenous nitrate vasodilator therapy or alternative interventions.

The aims of the study are:

1. To monitor the changes in concentration of cardiac biomarkers, VAS dyspnoea score and cardiac output before and after treatment of furosemide, isosorbide dinitrate or both.
2. To investigate whether the changes in concentration of cardiac biomarkers, VAS dyspnoea score and cardiac output before and after treatment is associated with the change in length of hospital stay.
3. To investigate whether combination treatment with intravenous furosemide and isosorbide dinitrate in patients with HF reduces VAS dyspnoea score, in-hospital mortality, length of hospital stay and number of readmission to a higher extend than do either medication alone.
4. To evaluate the prognostic values of novel cardiac biomarkers on 7-day, 14-day, 30-day and 6-month mortality and readmission.

Design:

This single-blinded randomized controlled study will be conducted in the Prince of Wales Hospital in Hong Kong.

Setting and Subjects:

Patients with dyspnoea will be screened and recruited from adult patients attending the emergency department at the Prince of Wales Hospital.

Interventions:

Patients with acute decompensated heart failure will be randomly treated with intravenous furosemide, isosorbide dinitrate or both. Level of dyspnoea, multi-biomarker and haemodynamic parameters will be measured before and after treatment.

Outcomes:

The primary outcome is the change in VAS dyspnoea score after treatment of furosemide, isosorbide dinitrate or both. The secondary outcomes are the changes in concentration of biomarkers and cardiac output, the number of in-hospital mortality, length of hospital stay, 7-day and 30-day and 6-month mortality and readmission.

DETAILED DESCRIPTION:
Definitions:

Heart failure can be defined as an abnormality of cardiac structure or function leading to failure of the heart to deliver oxygen at a rate commensurate with the requirements of the metabolizing tissues, despite normal filling pressures (or only at the expense of increased filling pressures).

Acute decompensated Heart Failure (ADHF), is defined according to Framingham criteria as a change in symptoms and signs in the context of heart failure. For this study we define this as an acute change in symptoms and signs within the previous 24 hours.

In the New York Heart Association classification (NYHA), Class I: no limitation is experienced in any activities; there are no symptoms from ordinary activities.; Class II: slight, mild limitation of activity; the patient is comfortable at rest or with mild exertion.; Class III: marked limitation of any activity; the patient is comfortable only at rest.; Class IV: any physical activity brings on discomfort and symptoms occur at rest.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with increased dyspnoea within the previous 24 hours
* Diagnosed as heart failure by physician

Exclusion Criteria:

* Women with known or suspected pregnancy; myocardial infarction or cardiac surgery within the previous three months;
* Oxygen saturation of less than 85% on room air;
* Respiratory rate greater than 30 breaths/min;
* pH<7.35; systolic blood pressure < 110 bpm;
* Current treatment with oral nitrates in excess of 40 mg daily;
* Current treatment with oral furosemide in excess of 80 mg daily;
* Previous adverse reaction to the study drugs;
* Requirement of noninvasive ventilation;
* Severe renal failure (creatinine >200 µmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
The change in VAS dyspnoea score after randomized treatment | 24 hour after recruitment
  Patients will be asked to indicate their status of dyspnoea using a visual analogue scale (VAS). They will be asked to make a mark on a 100 mm uncalibrated horizontal line in sitting (patients head at ≥ 600 relative to horizontal) and supine positions. The mark will be converted to a score (0-100 points) by measuring the distance from the left end. A VAS dyspnoea score of 0 corresponds to the patient's subjective feeling of "I can breathe normally" and a score of 100 represent to "I cannot breathe at all".

SECONDARY OUTCOMES:
The changes in concentration of biomarkers (including BNP, NTproBNP, NGAL, hs-CRP and ST2) after randomized treatment | 24 hour after recruitment
  5mL venous blood will be collected and applied to BNP, NTproBNP, NGAL and hs-CRP rapid test at baseline, 3 hours and 24 hours after randomized treatment at ED. The remaining blood will be centrifuged and stored at -20oC for ST2 measurement.
The changes in volume of blood pumped by the ventricle per minute (cardiac output) after randomized treatment | 24 hour after recruitment
  The cardiac output will be measured using an ultrasonic cardiac output monitor at baseline, 3 hours and 24 hours after randomized treatment at ED.
The number of in-hospital mortality | An average of 5 days
Number of day stayed in hospital | An average of 5 days
Number of mortality and readmission at 7-day, 14-day, 30-day and 6-month | 6-month after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Graham, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong